CLINICAL TRIAL: NCT06096701
Title: Use of a Cloud-connected Remote Blood Pressure Monitoring Program During the Postpartum Period for Hypertensive Women
Acronym: BP-ME
Status: Recruiting | Type: Observational
Sponsor: University of South Carolina (Other)
Collaborators: Prisma Health-Midlands (Other)
Responsible Party: Principal Investigator, Nansi Boghossian, Associate Professor, University of South Carolina
Other Study IDs: 2085188
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-03

CONDITIONS: Hypertensive Disorder
Keywords: Preeclampsia; Gestational hypertension; Eclampsia; Chronic hypertension
MeSH Terms: conditions — Hypertension; Pre-Eclampsia; Hypertension, Pregnancy-Induced; Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention: Intervention group will receive blood pressure (BP) cuffs. The BP cuff is connected in a Health Insurance Portability and Accountability Act-compliant fashion to the patient's medical record, allowing for documentation and communication with the nurse and the care team. Alerts are triggered if a patient has not checked her BP for 3 days or when readings fall outside a specific threshold (high or low BP alerts). Based on these alerts, the nurse follows up with these patients and reminds them to take a reading. The nurse will also notify participants with elevated BP values to repeat their BP and will contact the participants by phone to discuss symptoms and antihypertensive medications. Patients will be managed based on a clinical algorithm for initiation of antihypertensive medications without the need for an outpatient visit if considered appropriate by the clinical provider.
  Interventions: Device: Blood pressure cuff
- Historical or Concurrent controls: Individuals who had hypertensive disorders during pregnancy but who did not receive the BP cuffs will serve as the control group.

INTERVENTIONS:
Device: Blood pressure cuff — The BP cuff is connected in a Health Insurance Portability and Accountability Act-compliant fashion to the patient's medical record, allowing for documentation and communication with the nurse and the care team. Alerts are triggered if a patient has not checked her BP for 3 days or when readings fall outside a specific threshold (high or low BP alerts). Based on these alerts, the nurse follows up with these patients and reminds them to take a reading. The nurse will also notify participants with elevated BP values to repeat their BP and will contact the participants by phone to discuss symptoms and antihypertensive medications. Patients will be managed based on a clinical algorithm for initiation of antihypertensive medications without the need for an outpatient visit if considered appropriate by the clinical provider.
  Groups: Intervention

SUMMARY:
Hypertensive disorders (HD), including preeclampsia, gestational hypertension, chronic hypertension, and chronic hypertension with superimposed preeclampsia, affect around 10-20% of pregnant women in the United States and are significantly associated with maternal mortality and morbidity, particularly in the postpartum period. The prevalence of HD is on the rise in the United States and has increased from 13% in 2017 to 16% in 2019 owing to an increase in advanced maternal age, obesity, and diabetes. There are major racial disparities in HD and subsequent maternal mortality and morbidity. HD affect more than 1 in 5 delivery hospitalizations of Black women. Black women with HD are also more likely than white women with HD to have more adverse postpartum blood pressure trajectories which leads to a higher incidence of hypertension related hospital readmissions (readmission for hypertension during the first 6-weeks postpartum: 16.9% among Black women vs. 9.5% among white women, p=0.02) and cardiovascular-related adverse events. However, most of the management recommendations have been centered around blood pressure targets during the antepartum period with significantly less attention paid to the postpartum period despite evidence showing that hypertensive disorders are the most common reason for postpartum readmissions and are associated with increased maternal mortality and morbidity and a significant cost burden.

DETAILED DESCRIPTION:
Hypertensive disorders (HD), including preeclampsia, gestational hypertension, chronic hypertension, and chronic hypertension with superimposed preeclampsia, affect around 10-20% of pregnant women in the United States and are significantly associated with maternal mortality and morbidity, particularly in the postpartum period. The prevalence of HD is on the rise in the United States and has increased from 13% in 2017 to 16% in 2019 owing to an increase in advanced maternal age, obesity, and diabetes. There are major racial disparities in HD and subsequent maternal mortality and morbidity. HD affect more than 1 in 5 delivery hospitalizations of Black women. Black women with HD are also more likely than white women with HD to have more adverse postpartum blood pressure trajectories which leads to a higher incidence of hypertension related hospital readmissions (readmission for hypertension during the first 6-weeks postpartum: 16.9% among Black women vs. 9.5% among white women, p=0.02) and cardiovascular-related adverse events. However, most of the management recommendations have been centered around blood pressure targets during the antepartum period with significantly less attention paid to the postpartum period despite evidence showing that hypertensive disorders are the most common reason for postpartum readmissions and are associated with increased maternal mortality and morbidity and a significant cost burden.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals with hypertensive disorders
* Speak English
* At least 18 years old
* Medicaid coverage
* Between 20 weeks of pregnancy and 2 weeks postpartum
* Postpartum admission at Prisma Health Richland with hypertensive disorder within 2 weeks postpartum

Exclusion Criteria:

* Not planning to deliver at Prisma Health Richland
* Less than 20 weeks of pregnancy
* More than 2 weeks postpartum

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals who will deliver at Prisma Health Richland.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Blood pressure ascertainment | First 6 weeks postpartum
  BP ascertainment i.e., percent of patients submitting at least one BP value, the average number of unique BP measures per patient during the first six-weeks postpartum, and percent of patients continuing the program beyond 3 weeks postpartum.

SECONDARY OUTCOMES:
Percent of patients attending an in-person postpartum visit | First 8 weeks postpartum
Percent of patients readmitted to the hospital through 12 months postpartum | 12 months postpartum
Survey assessing patient's acceptability and satisfaction with the BP monitoring program | First 8 weeks postpartum
  The survey questions will include comfort with the technology and satisfaction with the BP monitoring program. All survey items will be assessed using a 5-item Likert scale (score of 1-strong disagreement, 3-neutral, 5-strong agreement) and will be administered through the telehealth platform starting on day 35 of the program. Patients who do not complete the survey will be contacted to complete it by phone or at their postpartum visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Prisma Health Richland, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No